CLINICAL TRIAL: NCT01891760
Title: A Prospective, Multi-center, Longitudinal, Cohort Study of Dermagraft in Subjects With Venous Leg Ulcers: A Long-term Follow-up to the DEVO-Trial
Brief Title: Long-Term Follow-Up to the DEVO Pivotal Trial of Dermagraft(R) to Treat Venous Leg Ulcers
Acronym: LTFU
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire Regenerative Medicine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABH-Dermagraft-001-09
Record Dates: First submitted 2013-06-28; First posted 2013-07-03 (Estimated); Last update posted 2013-08-21 (Estimated); Status verified 2013-08

CONDITIONS: Venous Leg Ulcer
MeSH Terms: conditions — Varicose Ulcer

ARMS (2):
- Treatment (Experimental): Dermagraft - Allogenic Neonatal Dermal Fibroblasts Seeded on poly(glycolide-co-L-lactide)(PGLLA)Scaffold
  Interventions: Device: Dermagraft
- Reference Therapy (Active Comparator): Profore - Four-layer compression bandaging therapy
  Interventions: Device: Profore

INTERVENTIONS:
Device: Dermagraft — Dermagraft treatment regimen of one application applied topically to the ulcer, weekly, for a maximum of 8 weeks (8 application maximum).
  Arms: Treatment
Device: Profore — Four-layer compression bandaging therapy.
  Arms: Reference Therapy

SUMMARY:
* Observe the long-term (1-year) outcomes of Dermagraft, compared with conventional treatment of four-layer compression bandaging therapy alone, in subjects who completed the ABH-Dermagraft-001-08 study.
* Study Hypothesis: N/A (Long-term follow-up study)

ELIGIBILITY:
Inclusion Criteria:

1. Subject has completed study ABH-Dermagraft-001-08
2. Subject understands study requirements
3. Subject is available to participate in the 1 year-long observational follow-up.

Exclusion Criteria:

1. Subject who withdrew or was terminated from ABH-Dermagraft-001-08 before completion
2. Subject is not available for the 1 year-long observational period.
3. Subject has any condition(s) which seriously compromises the subject's ability to complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2010-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
The incidence of study ulcer recurrence | 1 year

SECONDARY OUTCOMES:
Incidence of complete study ulcer healing | 1 year
Incidence of study ulcer infection-related events | 1 year
Time to study ulcer recurrence | 1 year
Change in ulcer size | 1 year
Time to study ulcer healing | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mollie Carter, MD, Study Director — Shire Regenerative Medicine
Locations (28):
- United States (12):
  - Carl T. Hayden VA Medical Center, Phoenix, Arizona
  - Hope Research Institute, Phoenix, Arizona
  - Dr. Jagpreet S. Mukker, Fresno, California
  - VA Northern California Health Care Sytem, Mather, California
  - North Amercian Center for Limb Preservation, New Haven, Connecticut
  - University of Miami Miller School of Medicine, Miami, Florida
  - Doctor's Research Network, South Miami, Florida
  - South Florida Wound Care Group, P.A., Tamarac, Florida
  - Covenant Wound Healing Center, Saginaw, Michigan
  - Advanced Foot & Ankle Center, Las Vegas, Nevada
  - Stony Brook University Medical Center, Stony Brook, New York
  - Saint Vincent Health Center, Erie, Pennsylvania
- East-Tallinn Central Hospital Department of Rheumatology, Tallinn, Estonia
- Germany (2):
  - Dermatologische Gemeinschaftspraxis Professor Dr. med W. Vanscheidt, Freiburg im Breisgau
  - Gemeinschaftspraxis Dres. Münter, Schiewe, Pohl Studienzentrum Dr. Münter, Hamburg
- Poland (6):
  - AKMed Medical Center, Department of Vascular Surgery, Krakow
  - Vascular Surgery, Tomasz Aleksiejew-Kleszczynski (Chirurgia Naczyn), Krakow
  - NZOZ "'Dermed" Medical Center (Centrum Medyczne Sp. z o.o., Lodz
  - "Medicos" Medical Center, Lublin
  - "NZOZ OPTI-MED Henryk Kaczmarek" Private Outpatient Clinic of Internal Medicine, Gastroenterology and Radiology, Nowy Sącz
  - NZOZ "Ars Medica" S.c. Wroclaw Health Centre (Wrocławskie Centrum Zdrowia), Wroclaw
- South Africa (6):
  - Lakeview Hospital, Benoni
  - Josha Research, Bloemfontein
  - Randles Road Medical Centre, Durban
  - GCT-Mercantile Clinical Trial Centre, Port Elizabeth
  - Cachetnied Medical Centre, Potchefstroom
  - Boland Ethical Research Group, Worcester
- Cardiff University Dept. of Wound Healing School of Medicine, Cardiff, United Kingdom

REFERENCES:
- See also: ClinicalTrials.gov registry for the Pivotal Trial of Dermagraft(R) to Treat Venous Leg Ulcers (DEVO) — http://clinicaltrials.gov/ct2/show/study/NCT00909870?term=DEVO&rank=1&view=record